CLINICAL TRIAL: NCT04296604
Title: Transcranial Direct Current Stimulation (tDCS) Neuromodulation of Executive Function Across Neuropsychiatric Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Chief of Division of Neuropsychiatry, Director of TMS Clinic, Director of Lab for Neuropsychiatry and Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P001428
Record Dates: First submitted 2020-02-28; First posted 2020-03-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury; Major Depressive Disorder; Bipolar Disorder; Schizophrenia; Attention Deficit Hyperactivity Disorder; Borderline Personality Disorder; Substance Use Disorders
Keywords: Transcranial Direct Current Stimulation; Executive Function
MeSH Terms: conditions — Brain Injuries, Traumatic; Depressive Disorder, Major; Bipolar Disorder; Schizophrenia; Attention Deficit Disorder with Hyperactivity; Borderline Personality Disorder; Substance-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (8):
- Traumatic Brain Injury (Experimental): This group consists of individuals diagnosed with traumatic brain injury. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Major Depressive Disorder (Experimental): This group consists of individuals diagnosed with major depressive disorder. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Bipolar Disorder (Experimental): This group consists of individuals diagnosed with bipolar disorder. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Schizophrenia (Experimental): This group consists of individuals diagnosed with schizophrenia. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Attention Deficit Hyperactivity Disorder (Experimental): This group consists of individuals diagnosed with attention deficit hyperactivity disorder. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Borderline Personality Disorder (Experimental): This group consists of individuals diagnosed with borderline personality disorder. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Substance Use Disorder (Experimental): This group consists of individuals diagnosed with substance use disorder. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation
- Healthy Controls (Active Comparator): This group consists of individuals diagnosed with healthy controls. This group will undergo three sessions of tDCS: two active sessions and one sham session. The order of the sessions is randomized.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, electrodes are applied on the scalp to transmit direct current at low current amplitudes.
  Other Names: tDCS

SUMMARY:
In the current study, the investigators aim to understand the role of transcranial direct current stimulation (tDCS) in improving executive function across neuropsychiatric populations known to have deficits in this cognitive domain.

DETAILED DESCRIPTION:
In the current study, the investigators aim to understand the role of transcranial direct current stimulation (tDCS) in improving executive function across neuropsychiatric populations known to have deficits in this cognitive domain. The investigators will select 8 relevant diagnostic categories: traumatic brain injury, major depressive disorder, bipolar disorder, schizophrenia, attention deficit hyperactivity disorder, borderline personality disorder and substance use disorder. The study will also include a cohort of healthy controls for comparison.

ELIGIBILITY:
Inclusion Criteria

1. Male and female outpatients 18-65 years of age
2. A diagnosis of traumatic brain injury, major depressive disorder, bipolar disorder, schizophrenia, attention deficit hyperactivity disorder, borderline personality disorder and substance use disorders meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.

Exclusion Criteria

1. Contraindication to tDCS: history or epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, shunts, pacemakers, pregnancy.
2. Active substance dependence (except for tobacco and cannabis).
3. Pregnant or nursing females.
4. Inability to participate in testing procedures.
5. Additional exclusion criteria for healthy controls:

   1. Diagnosis of psychiatric of neurological disorder
   2. Ongoing treatment with any psychotropic medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in N-Back Task | Baseline to Post-Treatment, 1 Week
  Working Memory Task

SECONDARY OUTCOMES:
Change in Flanker Task | Baseline to Post-Treatment, 1 Week
  Attention and Inhibitory Control Task
Change in Multi-Source Interference with International Affective Picture System Task | Baseline to Post-Treatment, 1 Week
  Cognitive Control During Emotional Regulation Task
Change in Delayed Discounting Task | Baseline to Post-Treatment, 1 Week
  Decision-Making Task
Change in Stop Signal Task | Baseline to Post-Treatment, 1 Week
  Ability to Inhibit a Response Task
Change in Iowa Gambling Task | Baseline to Post-Treatment, 1 Week
  Risk-Taking Task

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PhD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States